CLINICAL TRIAL: NCT04595305
Title: Septal Mapping And Resynchronisation Therapy- (SMART) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ABT-CIP-10291
Record Dates: First submitted 2020-08-02; First posted 2020-10-20 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Resynchronization Therapy; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm - Standard of Care (Other): Implantation of CRT-P or CRT-D for a clinical indication as per standard of care.
  Interventions: Device: Cardiac resynchronization therapy by CRT-P or CRT-D implantation

INTERVENTIONS:
Device: Cardiac resynchronization therapy by CRT-P or CRT-D implantation — Clinically indicated implantation of a CRT-P or CRT-D device as per standard of care
  Other Names: Cardiac resynchronization therapy

SUMMARY:
Normal heart function involves rhythmic contraction of all four chambers of the heart and this rhythm is maintained by the electrical wiring (conduction system) of the heart. Abnormality in this system results in either very slow or very fast heart rates leading to insufficient blood supply to the body due to inefficient pumping of the heart. cardiac resynchronization therapy pacemaker and cardiac resynchronization therapy defibrillator devices are used to synchronise heart function. The purpose of this study is not only to determine the pattern of electrical wiring of the heart and identify the variations seen in individuals with heart failure, but also, to explore the benefits of different types of pacing using CRT devices.

DETAILED DESCRIPTION:
Heart failure (HF) is an abnormality of cardiac structure or function leading to failure of the heart to deliver oxygen at the rate commensurate with the requirement of the patient or is able to do so only at the expense of elevated left ventricular filling pressures. European Society of Cardiology (ESC) 2016 guidelines defined HF as a syndrome in which patients have typical symptoms (e.g. breathlessness, swelling and fatigue) and signs (elevated jugular pressure, pulmonary crackles and displaced apex beat) resulting from an abnormality of cardiac structure or function. Patients with HF experience decreased exercise capacity, inability to perform activities of daily living, diminished quality of life, increased frequency of hospitalization and higher rates of mortality. HF is highly prevalent and affects approximately 26 million people worldwide with an estimated mortality of 50% within 5 years of diagnosis.1, 2 It remains a major threat to the public health system since more than 1 million patients are hospitalized with a primary diagnosis of HF annually, and, in western countries it is the most common cause of hospitalization in individuals >65 years of age.

Cardiac resynchronization therapy (CRT) using biventricular (BiV) pacing has been developed to restore synchrony in HF patients with delayed ventricular activation, predominantly of the left ventricle (LV). Studies have demonstrated that simultaneous or sequential BiV pacing restores the synchrony of contraction, reduces mitral regurgitation, and improves cardiac output. Several landmark clinical trials published in the past few years have provided compelling evidence that CRT can produce significant clinical benefits, including improvements in patients' HF symptoms, quality of life, hospitalization rates, and echocardiographic measures which confer a mortality benefit. Majority of patients show a benefit from CRT treatment however, up to 40% derive no improvement. In the MIRACLE study, 34% of patients did not demonstrate an improvement based on a clinical composite score (CCS) that combined all-cause mortality, HF hospitalization, New York Heart Association (NYHA) class and the Minnesota Living with Heart Failure Quality of Life Score. Birnie and Tang et al have summarized nonresponder rates from various clinical studies and the authors suggest that while most studies quote non-responder rates at 20-30% the true rate may be as high as 40-50%. They indicate that the inconsistencies might be largely due to the lack of standard definitions or methodologies to measure CRT response.

The precise mechanisms determining response are yet to be fully elucidated. It is generally believed that success is based on minimizing electrical activation times in the LV with a fusion between a left ventricular wavefront from a lead placed in the coronary sinus (CS) and a wavefront from a lead placed in the RV or an intrinsic wavefront.

The effects of different RV pacing sites have been varied in terms of their relationship to outcomes from CRT pacing. Initial smaller studies showed different outcomes between right ventricular apex (RVA) and outflow tract (RVOT) lead position, however further studies failed to demonstrate a benefit. Following this it was demonstrated that lead position initially believed to be septal were in fact antero-septal and that co-ordinated conduction would not be expected from these sites. Differing activation patterns have been demonstrated on Electroanatomic mapping (EAM) between intrinsic left bundle branch block (LBBB (circumferential)) and RV apical pacing (longitudinal). Another small study showed that RV lead placement at the site of latest activation during LV pacing improved acute haemodynamic measurements compared to standard RVA pacing, as did a true mid septal site compared to RVOT pacing - with the RV septum being the latest activated site during LV pacing when the CS lead was in the lateral vein.

LV septal activation has been proposed as a possible contributor to a successful response to CRT implantation. Trans-septal activation time has been shown in an animal model to correspond to the presence or absence of Heart failure when an LBBB is present, and successful acute haemodynamic response correlated to minimal epicardial activation time, LV endocardial pre-excitation and shortest QRS duration. Trans-septal conduction times have also been theorized to account for why QRS shortening with CRT is less than expected, however the degree to which this contributes is unknown.

Left ventricular total and septal scar have also been correlated to non-response to CRT. This would be expected to contribute to a longer trans-septal activation, as well as to local tissue strain measurement on echocardiography. Patterns of scar and their relationship to trans-septal activation times have not been documented. In the normal human heart up to three early endocardial sites have been documented and the location of scar relative to these sites and its effect is unknown. Earliest LV septal activation in LBBB heart failure patients may occur in mid septal regions suggesting activation of the LBB or outside of this region demonstrating direct trans-septal conduction, whether this correlates to CRT response is yet to be determined. Further evidence exists that there is a delay between electrical and mechanical activation of different cardiac segments (EMD), and that this is variable in the normal heart, as well as in the failing heart where it is further exacerbated between septal and lateral walls of the left ventricle. Reduction in total activation time may increase the total amount of myocardium recruited at any time point and that this may minimize EMD.

This single arm, non-randomized, open-label, multi-center, clinical investigation of 20 subjects is designed to characterize RV and LV septal activation patterns in CRT patients with various pacing configurations. The study will also assess the association of CRT response to septal activation patterns, septal scar and morphology of surface ECG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18 years of age or older, or of legal age to give informed consent specific to state and national law
* Subject must provide written informed consent prior to any clinical investigation related procedure
* Subjects who are undergoing implantation of an Abbott CRT-P or CRT-D device under standard indications
* Subjects are treated with optimal pharmacological therapy (as determined by the site principle investigator) for a minimum 4 weeks prior to procedure
* ECG showing Sinus Rhythm (SR)
* LBBB morphology with QRS duration >130ms
* Subject should be willing and able to comply with the prescribed follow-up schedule of evaluations.
* Female subjects of child-bearing potential should have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Exclusion Criteria:

* Subjects with a life expectancy less than the duration of the study
* Subjects with medical conditions that preclude the testing required for all patients by the study protocol or that otherwise limit study participation required for all patients
* Subjects with mechanical tricuspid or aortic heart valves
* Inaccessibility for follow-up at the study centre
* Unwillingness or inability to provide written informed consent
* Enrollment in, or intention to participate in, another clinical study during the course of this study excluding a registry
* Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Quantification of activation times (ms) of the RV and LV septum | During implant procedure
  Different pacing configurations such as LV-only pacing, biventricular pacing, and multipoint pacing will be used to quantify LV and RV septal activation time (ms).

SECONDARY OUTCOMES:
Quantification of the correlation coefficient relating changes in end-systolic volume (%) to the following variables: septal activation time (ms), septal scarring (% area), and ECG QRS duration (ms). | 12 months post-implant
  End-systolic volume (mL), which is an essential marker of cardiac function, may be dependent on septal activation time (ms), septal scarring (% area), and ECG QRS duration (ms). To test these relations, the correlation between changes in end-systolic volume in response to CRT and the aforementioned parameters will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: David O'Donnell, MD, FRACP, Principal Investigator — Fundacion GenesisCare
Locations (1):
- Abbott Medical Australia Pty Ltd, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No